CLINICAL TRIAL: NCT04688073
Title: Effect of Muscle Damage After Downhill Running on Postprandial Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chen-Kang Chang, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 201903HM011
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Nutritional and Metabolic Diseases; Lipemia
Keywords: triglyceride; non-esterified fatty acids; eccentric exercise; cardiovascular disease
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Hyperlipidemias; Cardiovascular Diseases | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Downhill running (Experimental): Running at 60% VO2max on -15% slope for 30 min on a treadmill
  Interventions: Behavioral: Exercise
- Level running (Experimental): Running at 60% VO2max on level surface for 30 min on a treadmill
  Interventions: Behavioral: Exercise
- Control (Placebo Comparator): Rest 30 min
  Interventions: Behavioral: Rest

INTERVENTIONS:
Behavioral: Exercise — Running
  Arms: Downhill running; Level running
Behavioral: Rest — sit and rest
  Arms: Control

SUMMARY:
All participants underwent three experimental trials, namely downhill running (DR), level running (LR), and the control (CON) in a cross-over design. Each trial lasted for 2 days. The participants were fed the same breakfast and lunch on day 1 in each trial. The participants arrived at the laboratory at 18:00 on day 1 and ran on the treadmill at 60% VO2max (downhill and level surface trials) or rested (CON trial) for 30 min. Subsequently, they were fed a standardized dinner (A meal box containing chicken, vegetables, and rice, 692 kcal, with 50% energy from carbohydrate, 32% from fat, and 18% from protein) within 20 min.

The participants returned to the laboratory at 07:30 on day 2 after an overnight fast. After baseline blood and gas samples were collected, the participants were fed a high-fat meal that included cereal, white bread, whipping cream, cheese, and butter. The high-fat meal provided fat 1.2 g/kg (65% energy), carbohydrate 1.1 g/kg (27% energy), protein 0.33 g/kg (8% energy), and 16.5 kcal/kg.

A 10-mL blood sample was collected from a forearm vein into nonheparinized tubes before and immediately after exercise or rest on day 1. On day 2, postprandial blood samples were collected from forearm veins into nonheparinized tubes by using an indwelling venous needle and a three-way stopcock. A 10-mL blood sample was collected before (0 h) and 0.5, 1, 2, 3, 4, 5, and 6 h after the high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy, had not engaged in regular exercise or received any medication in the past 6 months

Exclusion Criteria:

* history of cardiovascular disease, hypertension, hyperlipidemia, diabetes, atherosclerosis, or osteoporosis, free of any musculoskeletal injury during the study

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
TG AUC | 6 hours
  area under the curve for serum triglyceride concentrations within 6 hours after the high-fat meal

SECONDARY OUTCOMES:
NEFA AUC | 6 hours
  area under the curve for serum non-esterified fatty acid concentrations within 6 hours after the high-fat meal

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No